CLINICAL TRIAL: NCT00674323
Title: A Multicentre, Randomized, Double Masked, Exploratory, Indocyanine Green Angiography (ICGA) Guided Study of 6 Months Duration to Compare the Safety and Effect on Polyp Regression of Verteporfin Photodynamic Therapy (PDT) Alone or Added to Ranibizumab in Patients With Symptomatic Macular Polypoidal Choroidal Vasculopathy
Brief Title: Efficacy and Safety of Verteporfin Added to Ranibizumab in the Treatment of Symptomatic Macular Polypoidal Choroidal Vasculopathy
Acronym: PCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBPD952A2209
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal choroidal vasculopathy; PCV; Age-related macular degeneration (AMD) variant; vision; polyps; indocyanine green angiography; verteporfin; ranibizumab; photodynamic therapy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Macular Degeneration; Polyps | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Verteporfin and Ranibizumab (Experimental): Photodynamic therapy with verteporfin in combination with ranibizumab injection. Patients received one treatment at baseline with verteporfin photodynamic therapy (PDT) in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab intravitreal injection on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on indocyanine green angiography (ICGA), and assessment of fluorescein angiograms and visual acuity.
  Interventions: Drug: Verteporfin Photodynamic Therapy; Drug: Ranibizumab
- Verteporfin monotherapy (Active Comparator): Patients received one treatment at baseline with verteporfin photodynamic therapy in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab placebo (sham intravitreal injection) on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on indocyanine green angiography (ICGA), and assessment of fluorescein angiograms and visual acuity.
  Interventions: Drug: Verteporfin Photodynamic Therapy
- Ranibizumab monotherapy (Active Comparator): Patients received one treatment at baseline with verteporfin placebo (with sham photodynamic therapy) in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab intravitreal injection on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on indocyanine green angiography (ICGA), and assessment of fluorescein angiograms and visual acuity.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Verteporfin Photodynamic Therapy — After a 10-minute intravenous infusion of verteporfin at a dose of 6 mg/m^2 body surface area, light application of 50 J/cm^2 to the study eye was begun 15 minutes after the start of infusion.
  Other Names: Visudyne
  Arms: Verteporfin and Ranibizumab; Verteporfin monotherapy
Drug: Ranibizumab — Ranibizumab at dose of 0.5 mg administered as an intravitreal injection.
  Other Names: Lucentis
  Arms: Ranibizumab monotherapy; Verteporfin and Ranibizumab

SUMMARY:
This study aims to compare the efficacy of ranibizumab and verteporfin PDT combination treatment and verteporfin PDT monotherapy vs.ranibizumab monotherapy alone in achieving complete regression of polyps in patients with symptomatic macular polypoidal choroidal vasculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent before any assessment is performed.
* Male or Female patients ≥18 yrs of age
* Patients willing and able to comply with all study procedures

Inclusion criteria for study eye:

* BCVA letter score between 73-24 (approximately 20/40 to 20/320 Snellen equivalent) using ETDRS visual acuity chart measured at 4 meters
* PCV diagnosis confirmed by Central Reading Center
* Greatest Linear Dimension (GLD) of the total lesion area < 5400 µm (~9 Macular Photocoagulation Study Disc Areas)

Exclusion Criteria:

* Women of child-bearing potential who are not using one or more reliable contraception methods
* Pregnant or nursing (lactating) women
* History of hypersensitivity or allergy to fluorescein or indocyanine green (ICG), clinically significant drug allergy or known hypersensitivity to therapeutic or diagnostic protein products, or to any of the study drugs or their components
* Patient with history of porphyria
* Systemic medications known to be toxic to the lens, retina, or optic nerve
* History of which might affect the interpretation of the results of the study, or renders the patient at high risk from treatment complications
* Use of other investigational drugs within 30 days of randomization

Exclusion criteria for study eye:

* Concomitant conditions/diseases:
* Presence of angioid streaks, macular fibrosis, presumed ocular histoplasmosis syndrome, pathologic myopia (-8 Diopters or more)
* Active ocular inflammation or infection
* Uncontrolled glaucoma
* Ocular disorders that may confound interpretation of study results

Prior Ocular treatment:

* Prior Verteporfin PDT, external-beam radiation, laser photocoagulation, macular surgery, or transpupillary thermotherapy
* Prior local treatment with Pegaptanib, Ranibizumab, Bevacizumab or other anti-angiogenic compound or any investigational treatment in both eyes or systemic use of bevacizumab within 90 days prior to randomization
* History of intraocular surgery including pars plana vitrectomy and intraocular hemorrhage displacement is not allowed with the exception of uncomplicated cataract surgery that is allowed within 60 days prior to screening
* Ocular conditions that required chronic concomitant therapy within 90 days prior to randomization with topical, ocular, or systemically administered corticosteroids or any herbal medication known to contain steroid-like components

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis
Locations (5):
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Bangkok, Thailand

REFERENCES:
- [Derived] Tan CS, Ngo WK, Chen JP, Tan NW, Lim TH; EVEREST Study Group. EVEREST study report 2: imaging and grading protocol, and baseline characteristics of a randomised controlled trial of polypoidal choroidal vasculopathy. Br J Ophthalmol. 2015 May;99(5):624-8. doi: 10.1136/bjophthalmol-2014-305674. Epub 2015 Mar 10. PMID 25758601
- [Derived] Koh A, Lee WK, Chen LJ, Chen SJ, Hashad Y, Kim H, Lai TY, Pilz S, Ruamviboonsuk P, Tokaji E, Weisberger A, Lim TH. EVEREST study: efficacy and safety of verteporfin photodynamic therapy in combination with ranibizumab or alone versus ranibizumab monotherapy in patients with symptomatic macular polypoidal choroidal vasculopathy. Retina. 2012 Sep;32(8):1453-64. doi: 10.1097/IAE.0b013e31824f91e8. PMID 22426346

RESULTS

PARTICIPANT FLOW:
Groups:
- Verteporfin and Ranibizumab: Patients received one treatment at baseline with verteporfin photodynamic therapy (PDT) in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab intravitreal injection on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on indocyanine green angiography (ICGA), and assessment of fluorescein angiograms and visual acuity.
Period: Overall Study
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Started | 19 | 21 | 21
Completed | 18 | 20 | 21
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy | Total
Number analyzed (Participants) | 19 | 21 | 21 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.30) | 62.2 (9.77) | 69.3 (8.27) | 65.1 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 20
  Male | 11 | 15 | 15 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Regression (CR) of Polyps Measured by Indocyanine Green Angiography (ICGA)
Description: Indocyanine green angiography (ICGA) assessments were performed using the Heidelberg Retinal Angiography 2 (HRA2) machine to measure the Total Lesion Area and the degree of polyp regression. Complete regression was defined as no polyps seen on the imaging.
Time Frame: Month 6
Population: Full Analysis Set (FAS) included all patients randomized that received at least 1 application of study drug and had at least 1 post-baseline assessment of ICGA. Last Observation Carried Forward (LOCF) was utilized.
Measure: Number; unit: Participants
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Number analyzed (Participants) | 18 | 21 | 21
Participants | 14 | 15 | 6

2. Secondary Outcome: Number of Participants With at Least One Complete Polyp Regression During 6 Months Assessed by ICGA
Description: as for outcome 1
Time Frame: Baseline through end of study (6 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Number analyzed (Participants) | 18 | 21 | 21
Participants | 15 | 18 | 9

3. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness Measured by Optic Coherence Tomography (OCT)
Description: High resolution 6 meridian scans were performed to measure central retinal thickness.
Time Frame: Baseline and Month 6
Population: Full Analysis Set (FAS) included all patients randomized that received at least 1 application of study drug and had at least 1 post-baseline assessment of ICGA. LOCF was utilized.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Number analyzed (Participants) | 18 | 21 | 21
micrometers
  Baseline | 324.1 (112.72) | 285.3 (105.64) | 268.5 (97.84)
  Change from Baseline at month 6 | -145.6 (118.97) | -98.1 (104.33) | -65.7 (114.32)

4. Secondary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) of the Study Eye at Month 6
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increase in the VA score indicates improvement in visual acuity.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Number analyzed (Participants) | 18 | 21 | 21
Letters
  Baseline | 59.8 (16.21) | 57.2 (12.76) | 49.0 (18.05)
  Change from Baseline at Month 6 | 10.9 (10.92) | 7.5 (10.65) | 9.2 (12.39)

ADVERSE EVENTS:
Groups:
- Verteporfin and Ranibizumab: Patients received one treatment at baseline with verteporfin photodynamic therapy in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab intravitreal injection on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on ICGA, and assessment of fluorescein angiograms and visual acuity.
- Verteporfin Monotherapy: Patients received one treatment at baseline with verteporfin photodynamic therapy in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab placebo (sham intravitreal injection) on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on ICGA, and assessment of fluorescein angiograms and visual acuity.
- Ranibizumab Monotherapy: Patients received one treatment at baseline with verteporfin placebo (with sham photodynamic therapy) in the study eye and thereafter based on re-treatment criteria at intervals of at least 90 days. Within 1-24 hours, patients also received Ranibizumab intravitreal injection on Day 1 and at Month 1 and 2 and thereafter according to the re-treatment criteria at intervals of at least 30 days through Day 150. From month 3 onward, re-treatments were determined based on study-specific re-treatment criteria that included evaluation of polyp progression on ICGA, and assessment of fluorescein angiograms and visual acuity.
Arm/Group | Verteporfin and Ranibizumab | Verteporfin Monotherapy | Ranibizumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/21 | 2/21
Other Adverse Events (participants affected / at risk) | 8/19 | 9/21 | 4/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin and Ranibizumab (N=19) | Verteporfin Monotherapy (N=21) | Ranibizumab Monotherapy (N=21)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin and Ranibizumab (N=19) | Verteporfin Monotherapy (N=21) | Ranibizumab Monotherapy (N=21)
Conjunctival hyperaemia (Study eye) (Eye disorders) | 1 | 0 | 0
Dry eye (Study eye) (Eye disorders) | 1 | 1 | 0
Macular oedema (Study eye) (Eye disorders) | 1 | 0 | 0
Polypoidal choroidal vasculopathy (Fellow eye) (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 2 | 3 | 0
Visual impairment (Study eye) (Eye disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 0
Macular scar (Study eye) (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood pressure increased (Investigations) | 1 | 1 | 1
Intraocular pressure increased (Study eye) (Investigations) | 1 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.